CLINICAL TRIAL: NCT03613493
Title: Acceptability of HPV Self-sampling Tools for Cervical Cancer Prevention in Jamaican Women: A Theory-based Approach to Culturally-tailored Message Design
Brief Title: Acceptability of Human Papillomavirus (HPV) Self-sampling Tools for Cervical Cancer Prevention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Budgetary and Timing Constraints
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Susan Morgan, Associate Provost for Research Development and Strategy, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 20180033
Record Dates: First submitted 2018-06-17; First posted 2018-08-03 (Actual); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Cervical Cancer
Keywords: HPV; self-sampling; culture; message design; health communication; Jamaica
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- HPV self-sampling kit + Interview (Other): Participants will receive an HPV self-sampling kit to screen for HPV and then are interviewed about their experience using the tool.
  Interventions: Diagnostic Test: HPV self-sampling kit; Behavioral: Interview
- Culturally-targeted Fear appeal message HPV self-sampling kit (Experimental): Participants will receive an HPV self-sampling kit to screen for HPV, accompanied by a culturally-targeted fear appeal message
  Interventions: Diagnostic Test: HPV self-sampling kit; Behavioral: Culturally-targeted Fear Appeal Message
- Fear appeal message HPV self-sampling kit (Experimental): Participants will receive an HPV self-sampling kit to screen for HPV, accompanied by a culturally-targeted fear appeal message
  Interventions: Diagnostic Test: HPV self-sampling kit; Behavioral: Fear Appeal Message
- HPV self-sampling kit (Active Comparator): Participants will receive an HPV self-sampling kit to screen for HPV
  Interventions: Diagnostic Test: HPV self-sampling kit

INTERVENTIONS:
Diagnostic Test: HPV self-sampling kit — The HPV self-sampler kit will include the collection swab and the vial for collecting and storing the specimen, and an instructional sheet that visually depicts the steps for self-sampling.
Behavioral: Culturally-targeted Fear Appeal Message — Participants will receive culturally-targeted and fear appeal messages in a graphically designed kit.
  Arms: Culturally-targeted Fear appeal message HPV self-sampling kit
Behavioral: Fear Appeal Message — Participants will receive fear appeal messages (only) in a graphically designed kit.
  Arms: Fear appeal message HPV self-sampling kit
Behavioral: Interview — Participants will be interviewed about experiences using the self-sampling tool (qualitative).
  Arms: HPV self-sampling kit + Interview

SUMMARY:
The proposed study aims to increase HPV screening behaviors in Jamaican women by examining the acceptability of HPV Deoxyribonucleic Acid (DNA) self-sampling tools, and to determine the most culturally appropriate and effective message design for promoting such a tool in this context.

ELIGIBILITY:
Inclusion Criteria:

* Jamaican women, aged 30 to 65.

Exclusion Criteria:

* Women who report having had a hysterectomy,
* have had a history of cervical cancer,
* Women who are currently up-to-date on cervical cancer screening (have had a Pap in the last 3 years or have had a Pap smear/HPV co-test within the past 5 years),
* Adults unable to consent, children, pregnant women and prisoners.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Morgan, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HPV Self-sampling Kit + Interview | Culturally-targeted Fear Appeal Message HPV Self-sampling Kit | Fear Appeal Message HPV Self-sampling Kit | HPV Self-sampling Kit
Started | 10 | 75 | 0 | 90
Enrollment Criteria Met | 10 | 74 | 0 | 89
Completed | 10 | 73 | 0 | 83
Not Completed | 0 | 2 | 0 | 7

BASELINE CHARACTERISTICS:
Population: Due to budgetary constraints, participants were not enrolled into the Fear Appeal HPV self-sampler kit arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | HPV Self-sampling Kit + Interview | Culturally-targeted Fear Appeal Message HPV Self-sampling Kit | Fear Appeal Message HPV Self-sampling Kit | HPV Self-sampling Kit | Total
Number analyzed (Participants) | 10 | 74 | 0 | 89 | 173
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.40 (9.442) | 45.01 (9.099) |  | 41.09 (10.222) | 44.50 (9.587)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 74 | 0 | 89 | 173
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 74 | 0 | 89 | 173
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 74 | 0 | 89 | 173
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Prior pap test experience [Number; unit: participants] | 7 | 64 |  | 72 | 143

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Used and Returned Their Self-sampler Kit.
Description: Number of participants that used and returned their self-sampler kit was evaluated.
Time Frame: 2 weeks
Population: Data was not collected for the fear appeal message HPV self-sampling condition due to lack of funding.
Measure: Count of Participants; unit: Participants
Arm/Group | Culturally-targeted Fear Appeal Message HPV Self-sampling Kit | Fear Appeal Message HPV Self-sampling Kit | HPV Self-sampling Kit | HPV Self-sampling Kit + Interview
Number analyzed (Participants) | 74 | 0 | 89 | 10
Participants | 73 |  | 83 | 10

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | HPV Self-sampling Kit + Interview | Culturally-targeted Fear Appeal Message HPV Self-sampling Kit | HPV Self-sampling Kit
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/74 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/74 | 0/89
Other Adverse Events (participants affected / at risk) | 0/10 | 0/74 | 0/89

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/93/NCT03613493/Prot_SAP_000.pdf